CLINICAL TRIAL: NCT04472065
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of a Probiotic Dietary Supplement on the Gut Microbiome, Oxytocin Levels, Socio-emotional Functioning, and Well-being in Mother-Infant Dyads
Brief Title: Study of Probiotic Use After Childbirth in Relation to Emotional Well-Being
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Austen Lawson (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Austen Lawson, Elizabeth A. Lawson, M.D., M.M.Sc., Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2020P000562
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Mental Health Wellness
Keywords: Gut microbiome; Postpartum depression; Oxytocin; Socio-emotional functioning; Probiotic
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Expectant mothers who meet eligibility criteria will be randomized 1:1, stratified by C-section or vaginal delivery, to either the probiotic dietary supplement group or the placebo group and will be blinded to treatment assignment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be performed by the unblinded study pharmacist. All study staff will be blinded to treatment assignment. The infant will be assigned to the same group as their mother.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subjects receiving Probiotic Dietary Supplement (Active Comparator)
  Interventions: Dietary Supplement: Lactobacillus reuteri
- Subjects receiving Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — 1 chewable tablet of probiotic dietary supplement (200 million CFU of L. reuteri DSM 17938 and ATCC PTA 6475) consumed once per day orally for 6 weeks beginning at Baseline (between 1 to 3 days postpartum) to 6 weeks postpartum.
  Arms: Subjects receiving Probiotic Dietary Supplement
Other: Placebo — 1 chewable placebo tablet containing all the same ingredients except L. reuteri (DSM 17938 and ATCC PTA 6475) consumed once per day orally for 6 weeks beginning at Baseline (between 1 to 3 days postpartum) to 6 weeks postpartum.
  Arms: Subjects receiving Placebo

SUMMARY:
Researchers at Massachusetts General Hospital are interested in learning more about the neurobiology of well-being in new mothers and novel ways to support them during their transition to parenthood. This study aims to evaluate well-being in new mothers and their infant and the impact of a probiotic dietary supplement on the gut microbiome. This study hopes to help improve the existing knowledge of maternal postnatal health.

ELIGIBILITY:
Inclusion Criteria

1. Able and willing to give written informed consent
2. Expectant mothers with singleton infant or mothers who have recently given birth to a singleton infant
3. At least 18 years of age
4. At risk for postpartum depression as defined: a hx of depression and/or, a hx of postpartum depression and/or by a prenatal EPDS score ≥ 8

Exclusion Criteria:

1. Has active substance abuse in the past 6 months or a history of opioid use disorder
2. Has diabetes mellitus except for diet controlled gestational diabetes
3. Has uncontrolled thyroid disease
4. Has inflammatory gastrointestinal disease
5. Has active suicidal ideation
6. Has a history of psychosis
7. Has a history of an autism spectrum disorder
8. Plans to take other probiotics (other than study product) during study participation
9. Plans to take systemic hormonal contraception during study participation (Note: intra-uterine device is allowed)
10. Is receiving any systemically administered immunosuppressant medication on a chronic basis
11. Has a clinically significant or uncontrolled concomitant illness or condition that would put the subject at risk or jeopardize the objectives of the study
12. Has a contraindication, sensitivity, or known allergy to any ingredient of the study product
13. Is considered, in the opinion of the Principal Investigator (PI), to likely be a poor attendee or unlikely for any reason to be able to comply with the study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Coding Interactive Behavior (CIB) Negative Scale Score (range: 1-5; direction: Higher values indicate worse maternal responses) in the probiotic versus placebo group | 6 week
  Mother-infant bonding: Quantitative observational assessment of mother-infant bonding using the Child Interactive Behavior (CIB).

SECONDARY OUTCOMES:
Change in Toronto Alexithymia Scale (TAS-20) Total Score (range: 20-100; direction: lower scores indicate better socioemotional functioning) in the probiotic versus placebo group | Baseline to Week 6
Change in relative abundance of microbial taxa (operational taxonomic units) in fecal samples in the probiotic versus placebo group | Baseline to Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Lawson, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States